CLINICAL TRIAL: NCT05791604
Title: The Safety and Effectiveness Study of Prebiotics and Probiotics in the Intervention of Obesity in Children With Prader-Willi Syndrome
Brief Title: The Intervention of Obesity in Children With Prader-Willi Syndrome Using Prebiotics and Probiotics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PREPROPWS
Record Dates: First submitted 2023-03-06; First posted 2023-03-30 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi syndrome; Probiotics; Prebiotics
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Prebiotics; galactomannan; oligofructose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotics group (Experimental): Take probiotics during the study
  Interventions: Dietary Supplement: probiotics including B. lactis B420, B. lactis HN019, B. animalis Bb-12, L. rhamnosus GG
- Probiotics and prebiotics group (Experimental): Take probiotics and prebiotics during the study
  Interventions: Dietary Supplement: probiotics including B. lactis B420, B. lactis HN019, B. animalis Bb-12, L. rhamnosus GG; Dietary Supplement: Prebiotics with galactomannan and oligofructose
- Control group (No Intervention): Take placebo food during the study

INTERVENTIONS:
Dietary Supplement: probiotics including B. lactis B420, B. lactis HN019, B. animalis Bb-12, L. rhamnosus GG — Take probiotics, 2g each time, twice a day, for 12 weeks
  Arms: Probiotics and prebiotics group; Probiotics group
Dietary Supplement: Prebiotics with galactomannan and oligofructose — Take probiotics, 2g each time, twice a day, for 12 weeks Take prebiotics, 25g each time, twice a day, for 12 weeks
  Arms: Probiotics and prebiotics group

SUMMARY:
Prader-Willi syndrome (PWS) is a rare genetic disease, with hyperappetite and severe obesity. At present, there is no effective drugs and interventions to help control the appetite of PWS patients. More and more evidence has shown that gut microbiota is closely related to obesity. Probiotics and prebiotics can improve the structure of gut microbiota, thus improve blood lipid levels and other biochemical indicators of obese people. Therefore, this study intends to explore the effectiveness and safety of probiotics and prebiotics in controlling appetite and weight gain of PWS children.

DETAILED DESCRIPTION:
Prader-Willi syndrome (PWS) is a rare genetic disease, with hyperappetite and severe obesity. Morbid obesity and related complications caused by hyperappetite are the most common causes of poor prognosis and death in PWS. At present, there is no effective drugs and interventions to help control the appetite of PWS patients. At present, more and more evidence has shown that gut microbiota is closely related to obesity. Probiotics and prebiotics can improve the structure of gut microbiota, thus improve blood lipid levels and other biochemical indicators of obese people. Therefore, this study intends to explore the effectiveness and safety of probiotics and prebiotics in controlling appetite and weight gain of PWS children. Participants will be divided into three groups, receiving probiotics, probiotics+probiotics or placebo treatment, and observe the changes in body weight, the structure of gut microbiota and metabolic level.

ELIGIBILITY:
Inclusion Criteria:

* Pre-adolescent children with Prader Willi syndrome which were definitely diagnosed by gene testing.
* Consistent with the diagnostic criteria for obesity.
* Not participate in other research projects at present or three months before the research;
* Agree to participate in the test and obtain the consent of their parents; voluntarily be the subjects and sign the informed consent form.

Exclusion Criteria:

* Losing weight in ways other than the intervention measures of this project, such as taking weight loss drugs or known drugs that cause weight change;
* Use antibiotics within 1 month before the study and lasted for 3 days or more;
* Use probiotics within 1 month before the study and lasted for 3 days or more;
* Complicated with liver and renal insufficiency (alanine aminotransferase and serum creatinine indexes exceed 2 times the upper limit of the normal value set by the hospital);
* Have gastrointestinal diseases affecting food digestion and absorption (such as severe diarrhea, constipation, severe gastrointestinal inflammation, active gastrointestinal ulcer, acute cholecystitis, etc.); severe diarrhea refers to watery stool 3 or more times a day and lasts for 3 or more days. severe constipation refers to defecation 2 or less times a week with difficulty in defecation;
* Surgery was performed within 1 year before the study (except for appendicitis and hernia surgery);
* Have hepatitis B, active tuberculosis, AIDS and other infectious diseases;
* Those who are suffering from mental illness and are taking psychotropic drugs such as antidepressants.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Body mass index | 12 weeks
  Body mass index is calculated as weight (kg)/[Height (m)^2]. Weight and height will be combined to report BMI in kg/m^2.

SECONDARY OUTCOMES:
Body composition | 4 weeks and 12 weeks
  Body composition including body fat percentage will be measured through body composition meter.
The structure of gut microbiota | 4 weeks and 12 weeks
  The 16s rRNA genes of fecal samples were analyzed.
Height | 4 weeks and 12 weeks
  The height is accurate to 0.1cm.
Weight | 4 weeks and 12 weeks
  The weight is accurate to 0.1kg.
Waist circumference | 4 weeks and 12 weeks
  The waist circumference is accurate to 0.1cm.
Glycosylated hemoglobin level | 4 weeks and 12 weeks
  The glycosylated hemoglobin is accurate to 0.1%.
Fast triglyceride level | 4 weeks and 12 weeks
  The fast triglyceride level will be measured by IMMULITE 1000 (Siemens,Germany).
Fast total cholesterol level | 4 weeks and 12 weeks
  The fast total cholesterol level will be measured by IMMULITE 1000 (Siemens,Germany).
Fast low density lipoprotein level | 4 weeks and 12 weeks
  The fast low density lipoprotein level will be measured by IMMULITE 1000 (Siemens,Germany).
Fast high density lipoprotein level | 4 weeks and 12 weeks
  The fast high density lipoprotein level will be measured by IMMULITE 1000 (Siemens,Germany).
Defecation status | 4 weeks and 12 weeks
  Care givers describe the defecation status in the past 1 week, including the frequency, nature, and color.
Abdominal pain | 4 weeks and 12 weeks
  Care givers describe whether abdominal pain occurs, and if so, provide frequency.
Excessive flatulence | 4 weeks and 12 weeks
  Care givers describe whether excessive flatulence occurs, and if so, provide frequency.
Fast insulin level | 4 weeks and 12 weeks
  The fast insulin level will be measured by IMMULITE 1000 (Siemens,Germany).
Fast glucose level | 4 weeks and 12 weeks
  The fast glucose level is detected by fingertip blood with blood glucose meter.
Body mass index | 4 weeks
  Body mass index is calculated as weight (kg)/[Height (m)^2]. Weight and height will be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Lu, Dr, Study Director — Children's Hospitial of Fudan Univeristy
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
After applying to the researcher, the researcher will decide whether to share the data

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT05791604/Prot_SAP_ICF_000.pdf